CLINICAL TRIAL: NCT00267358
Title: Placebo Controlled, Randomized Safety and Efficacy Study of RC-1291 in Cancer Anorexia/Cachexia.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Helsinn Therapeutics (U.S.), Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: RC-1291-205
Record Dates: First submitted 2005-12-19; First posted 2005-12-20 (Estimated); Last update posted 2013-09-02 (Estimated); Status verified 2013-08

CONDITIONS: Cancer Cachexia

ARMS (2):
- RC-1291 HCl (Active Comparator): 50 mg
  Interventions: Drug: RC-1291 HCl
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RC-1291 HCl
  Arms: RC-1291 HCl
Drug: Placebo
  Arms: Placebo

SUMMARY:
Anorexia and cachexia are devastating complications in late-stage cancer patients and is strongly associated with mortality in these patients. Activation of Ghrelin receptors have been demonstrated to stimulate appetite. RC-1291 HCl, by virtue of its ghrelin like activity and Growth Hormone releasing effects may have a dual role in the reversal of cancer induced anorexia and cachexia. This placebo controlled study will evaluate the safety and efficacy of RC-1291 HCl in cancer patients with anorexia and cachexia.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling patients ≥ 18 years of age with incurable,histologically diagnosed cancer.
* Involuntary loss of body weight of ≥ 5 % within the past 6 months

Exclusion Criteria:

* Presently hospitalized or in a nursing care facility.
* Inability to increase food intake from secondary causes.
* Liver disease
* If female-pregnant, breast-feeding or of childbearing potential.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2005-11; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Body weight
Lean body mass
Functional performance

CONTACTS AND LOCATIONS:
Overall Officials: William Polvino, MD, Study Director — Helsinn Therapeutics (U.S.), Inc
Locations (19):
- United States (19):
  - Palo Verde Hematology Oncology Ltd., Glendale, Arizona
  - Comprehensive Blood & Cancer Center, Bakersfield, California
  - Pacific Oncology & Hematology Associates, Encinitas, California
  - Pacific Oncology and Hematology Associates, Encinitas, California
  - Advanced Medical Research Institute, Fresno, California
  - Kenmar Clinical Research, Los Angeles, California
  - Kenmar Research Institute, Los Angeles, California
  - Sant Chawla, Inc., Santa Monica, California
  - PAB Clinical Research, Brandon, Florida
  - Melbourne Internal Medicine Associates, Melbourne, Florida
  - Osler Medical, Inc./ Osler Clinical Research, Melbourne, Florida
  - Bay Area Oncology, Tampa, Florida
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Hematology Oncology Consultants, Inc., Columbus, Ohio
  - Charleston Cancer Center, Charleston, South Carolina
  - South Carolina Oncology Associates, Columbia, South Carolina
  - South Carolina Cancer Specialists, Hilton Head Island, South Carolina
  - University of Texas Medical Texas, Galveston, Texas
  - Multicare Health System, Tacoma, Washington

REFERENCES:
- [Derived] Garcia JM, Boccia RV, Graham CD, Yan Y, Duus EM, Allen S, Friend J. Anamorelin for patients with cancer cachexia: an integrated analysis of two phase 2, randomised, placebo-controlled, double-blind trials. Lancet Oncol. 2015 Jan;16(1):108-16. doi: 10.1016/S1470-2045(14)71154-4. Epub 2014 Dec 16. PMID 25524795